CLINICAL TRIAL: NCT04570462
Title: Application of Mild Hypothermia for COVID-19 Acute Respiratory Distress
Brief Title: Mild Hypothermia for COVID-19 ARDS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was opened at the close of the peak of COVID. At our institution, there are significantly less COVID patients admitted who qualify for the study
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Pey-Jen Yu, MD, Director, Clinical Research Programs, Department of Cardiovascular and Thoracic Surgery, North Shore University Hospital, Northwell Health, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 5.18.2020 Approved
Record Dates: First submitted 2020-07-21; First posted 2020-09-30 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2020-09

CONDITIONS: COVID19 ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm- Induction of Mild Hypothermia Protocol (Experimental): Determination of metabolic rate by the metabolic cart (noninvasive connection of the device to the ventilator for 20 minutes). Initiate hypothermia (established Northwell hypothermia status post cardiac arrest protocol) using the Arctic Sun. The Arctic Sun 5000® is set to a temperature of 34.5 C to lower the body temperature.
  Interventions: Other: Hypothermia Via Cooling Machine- Arctic Sun 5000

INTERVENTIONS:
Other: Hypothermia Via Cooling Machine- Arctic Sun 5000 — Initiate hypothermia using the Arctic Sun.The Arctic Sun 5000® is set to a temperature of 34.5 C to lower the body temperature.
  Duration of hypothermia will be 48 hours after which the subject will be rewarmed. Metabolic rate, or indirect Calorimetry, will be assessed at baseline, day 1 of hypothermia, day 2 of hypothermia before rewarming, and after full rewarming. CBC, basic metabolic profile, magnesium, phosphorus, coagulation profile, ABG, inflammatory markers would be drawn every 12 hours during hypothermia until subject has achieved full rewarming and once after full rewarming.
  The entire hypothermia procedure will last 48 hours. Acceptable rewarming range is a temperature of 36.5C to 37.5C. The subject body temperature rewarming is typically set over 6-8 hours. Therefore, the final 6-8 hours of the 48 hour time period is set to rewarm the subject.

SUMMARY:
Some patients with COVID have abnormally high carbon dioxide and low oxygen levels despite being on the ventilator. The hypothesis of the study is that the application of mild hypothermia to patients with COVID will decrease their metabolic rate and improve their oxygenation and carbon dioxide levels.

DETAILED DESCRIPTION:
A significant contributor to the morbidity and mortality from COVID-19 is from the abnormal carbon dioxide and oxygen levels in COVID-19 patients. Metabolic studies done on COVID-19 patients have shown that these patients have abnormally high metabolic rates. High metabolic rates results in increased carbon dioxide production and increased oxygen usage, both of which can result in high carbon dioxide and low oxygen levels. As some patients with severe COVID-19 continue to have high carbon dioxide levels and/or low oxygen levels despite being on the ventilator, it is hypothesized that decreasing the metabolic rate in these COVID-19 patients will help their oxygen and carbon dioxide levels. Mild hypothermia is currently used in comatose survivors of cardiac arrest to improve mortality and neurological outcomes. Mild hypothermia is also an effective way to reduce metabolic demand. The aim is to apply mild hypothermia to COVID-19 patients to decrease metabolic rate in order to improve their oxygen and carbon dioxide levels. Although the application for mild hypothermia has been widely adopted in some patient populations, it has never been applied in COVID-19 patients. If we can develop a strategy to help improve the oxygen and carbon dioxide levels in COVID-19 patients, it may lead to improvements in their overall outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form from Legally Authorized Representative.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or above
4. COVID positive
5. On mechanical ventilation with either: refractory respiratory acidosis (ph ≤ 7.20), hypercarbia (pCO2 ≥ 55 mmHg), refractory hypoxia (pO2/FIO2 <150), or plateau pressures >30

Exclusion Criteria:

1. Bleeding (active bleeding, platelets less than 50,000)
2. Uncontrolled cardiac arrhythmia
3. History of cryoglobulinemia, major trauma, pregnancy
4. Active non-COVID-19 infection that is not controlled with antibiotic or antifungal regimen

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic requirement during and after hypothermia | Every 12 hours through study completion an average of 4 days
  indirect calorimeter measurements (Kcal/day)

SECONDARY OUTCOMES:
Changes in oxygen requirements and levels during and after hypothermia | Every 12 hours through study completion, an average of 4 days
  ABG, PaO2 (mmHg)
length of intubation | through study completion, an average of 4 days
  number of hours intubated
Changes in carbon dioxide levels during and after hypothermia | Every 12 hours through study completion an average of 4 days
  measured by ABG, PaCO2 mmHg
does application of hypothermia reduce pro inflammatory response | through study completion an average of 4 days
  ESR (mm/hr)
does application of hypothermia reduce pro inflammatory response | through study completion an average of 4 days
  Ferritin (ng/ml)
does application of hypothermia reduce pro inflammatory response | through study completion an average of 4 days
  D Dimer (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT04570462/Prot_SAP_000.pdf